CLINICAL TRIAL: NCT00499811
Title: Phase I and Pharmacokinetic Study of Vorinostat for Solid Tumors and Lymphomas in Patients With Varying Degrees of Hepatic Dysfunction
Brief Title: Vorinostat in Treating Patients With Metastatic or Unresectable Solid Tumors or Lymphoma and Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00272; NCI-2009-00272 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-07-C-0228; CDR0000555102; PCI-UPCI 07-013; UPCI 07-013 (Other: University of Pittsburgh); 8057 (Other: CTEP); N01CM62208 (NIH); U01CA099168 (NIH); U01CA062505 (NIH); U01CA062491 (NIH); U01CA062487 (NIH); P30CA047904 (NIH)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Primary Central Nervous System Hodgkin Lymphoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Vorinostat

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Vorinostat (SAHA) will be administered as a single oral dose on day -6 for all patients. Blood samples are obtained periodically on day -6 for pharmacokinetic studies.
  One week later (day 1), the first course of oral vorinostat will be initiated on a continuous daily oral regimen. Each treatment course will consist of 21 days of therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Other: pharmacological study

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat in treating patients with metastatic or unresectable solid tumors or lymphoma and liver dysfunction. (closed for accrual as of 04/05/2010) Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Vorinostat may have different effects in patients who have changes in their liver function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the pharmacokinetic disposition of vorinostat (SAHA) in patients with metastatic or unresectable solid tumors or lymphoma and varying degrees of hepatic dysfunction.

II. Establish the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of vorinostat in groups of patients with varying degrees of hepatic dysfunction (mild, moderate, or severe).

SECONDARY OBJECTIVES:

I. Document the non-DLTs associated with administration of vorinostat in patients with hepatic dysfunction.

II. Determine the association of the Child-Pugh classification of hepatic dysfunction with the observed toxicities, plasma pharmacokinetics, and pharmacodynamics of vorinostat administration.

III. Document any antitumor activity associated with vorinostat treatment in patients enrolled on this study.

OUTLINE: This is a parallel-group, dose-escalation study. Patients are stratified according to level of hepatic dysfunction (normal vs mild vs moderate vs severe). (closed for accrual as of 04/05/2010)

PART I: Vorinostat (SAHA) will be administered as a single oral dose on day -6 for all patients. Blood samples are obtained periodically on day -6 for pharmacokinetic studies.

PART II: One week later (day 1), the first course of oral vorinostat will be initiated on a continuous daily oral regimen. Each treatment course will consist of 21 days of therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

Dose escalation will proceed within each hepatic dysfunction group (except in the normal group). Only dose-limiting toxicities (DLTs) that occur during the first cycle of treatment will be used to guide dose escalation. The maximum tolerated dose (MTD) is the highest dose at which no more than one instance of DLT is observed (among 6 patients treated). Once the MTD has been determined for a given hepatic dysfunction group, a maximum of 12 patients will be accrued to this dose level.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid malignancy or lymphoma that is metastatic or unresectable

  * Patients with a liver mass, elevated α-fetoprotein level (≥ 500 ng/mL), and positive serology for hepatitis consistent with a diagnosis of hepatocellular carcinoma will be eligible without the need for pathologic confirmation of the diagnosis
* Standard curative or palliative measures do not exist or are no longer effective

  * Patients who have not received any prior therapy for malignancy are also eligible if they are ineligible for standard therapy due to hepatic dysfunction
* Patients with abnormal liver function will be eligible

  * No distinction will be made between liver dysfunction due to metastases and liver dysfunction due to other causes
  * Patients with biliary obstruction for which a shunt has been placed are eligible, provided the shunt has been in place for at least 10 days prior to the first dose of vorinostat (SAHA) and liver function has stabilized

    * Two measurements at least 2 days apart that put the patient in the same hepatic dysfunction stratum will be accepted as evidence of stable hepatic function
  * No evidence of biliary sepsis
* Patients with gliomas or brain metastases who require corticosteroids or anticonvulsants must be on a stable dose of corticosteroids and seizure free for 1 month prior to study enrollment

  * Patients with known brain metastases should have had brain irradiation (whole brain or gamma knife) more than 4 weeks before starting protocol treatment
  * Patients with unstable or untreated (non-irradiated) brain metastases should be excluded
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* Life expectancy > 3 months
* Absolute neutrophil count > 1,500/mm^3
* Platelets ≥ 100,000/mm^3
* Creatinine within normal institutional limits OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV-positive patients without an AIDS-defining diagnosis who are not receiving agents with the potential for pharmacokinetic interactions with vorinostat may be eligible
* Able to take oral medications on a continuous basis
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No active hemolysis
* More than 3 weeks since prior chemotherapy or radiotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered

  * Patients who have been treated with agents that persist in the body for longer than 4 to 6 weeks (such as suramin) are ineligible during the elimination period for those agents
* More than 14 days since prior major surgery
* No prior vorinostat
* At least 2 weeks since prior valproic acid or other histone deacetylase inhibitors
* More than 4 weeks since other prior investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent therapy with enzyme-inducing anticonvulsants
* No concurrent prophylactic granulocyte growth factors during the first cycle of therapy
* No other concurrent investigational or commercial agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-06; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) variables corresponding to the disposition of vorinostat (SAHA) (Group 1) | Days -6 and 1 of course 1
  The Wilcoxon test will be used for PK data. Concentrations of vorinostat and 2 metabolites (vorinostat glucuronide and 4-anilino-4-oxobutanoic acid) will be quantitated with a liquid chromatography-electrospray ionization tandem mass spectrometric method that was developed and validated in our laboratory. Plasma concentration versus time data for vorinostat and metabolites will be analyzed non-compartmentally using the LaGrange function as implemented by the Lagran computer program.
MTD of vorinostat based on incidence of DLT | Up to 21 days
  The MTD is the highest dose at which no more than one instance of DLT is observed (among 6 patients treated). The MTDs determined in this study represent a simple summary of the relationship between the dose of vorinostat that can be administered with acceptable toxicity and a patient's level of liver dysfunction. Treatment-related events occurring during the first course of treatment are considered DLTs.

SECONDARY OUTCOMES:
Toxicity profile of vorinostat | Up to 4 weeks after completion of treatment
  Toxicities will be graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0. The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category, grade. Tabulations will be separate for each liver dysfunction group, and may also be separate for each dose level within a group, if appropriate. For grade 3-4 toxicity, analyses will utilize Fisher's exact test.
Clinical response rate | Up to 4 weeks after completion of treatment
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.
Child-Pugh classification and liver function test results | At baseline
  The Child-Pugh Classification and its association with toxicity and PK data will be studies in an exploratory analysis. For grade 3-4 toxicity, analyses will utilize Fisher's exact test; for PK data, the Wilcoxon test will be used. In addition, the correlation between the level(s) of liver dysfunction (bilirubin and/or synthetic (albumin), hepatocellular (bilirubin, ALT, AST) and/or ductal (gamma-GT, alkaline phosphatase) parameters and alterations in the PK of vorinostat will be evaluated with Spearman's test

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, Principal Investigator — University of Pittsburgh
Locations (11):
- United States (11):
  - City of Hope Medical Center, Duarte, California
  - University of Southern California, Los Angeles, California
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - National Institutes of Health, Bethesda, Maryland
  - Wayne State University-Karmanos Cancer Institute, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin